CLINICAL TRIAL: NCT06851637
Title: Reducing Symptoms of Depression, Stress and Anxiety and Enhancing Positive Mental Health: a Randomized-controlled Study of the Positive Emotions Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Lara Steinmann, Master of Science (M. Sc.) in Clinical Psychology, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PoET102
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Positive Emotions; Mental Health; Intervention (Training) Condition; Randomized Controlled Study; General Population (no Specific Condition or Disease)
Keywords: positive emotions; online intervention; positive psychology; randomized controlled study; intervention; general population
MeSH Terms: conditions — Psychological Well-Being; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PoET group (Experimental): Participants of this arm received the PoET online training within two sessions. They filled out a whole of three questionnaires.
  Interventions: Behavioral: PoET
- Control group (No Intervention): Participants did not receive any treatment initially, but were offered to participate in a later PoET training as compensation. They filled out a whole of three questionnaires.

INTERVENTIONS:
Behavioral: PoET — Participants in the PoET group completed two online training sessions (3 hours each) via Zoom. Group size was about 25-30 people. The sessions included the following positive psychology constructs: happiness, humour, optimism, loving kindness and gratitude on the first day, and hope, self-efficacy, meaningfulness, forgiveness and resilience on the second day.
  Arms: PoET group

SUMMARY:
Based on the results of the previously published paper "Positive Emotions Training (PoET) as an online intervention to improve mental health: a feasibility study" (Niemann et al., 2023) the goal of this study was to examine the effects of the "Positive Emotions Training" on mental health in a randomized-controlled study. Furthermore, possible predictors for the efficacy of PoET are to be explored.

Hypotheses:

1. It was hypothesized that participants receiving PoET would show a significant increase in positive mental health factors at the second assessment point (T2) at end of the second training day.
2. Furthermore, participants receiving PoET are to be expected to show a significant decrease in depression, anxiety and stress symptoms at T2.
3. It was hypothesized that the changes in mental health factors remain stable up to the last assessment point (T3) three month after the training.
4. Lastly, it was hypothesized that there would be no significant changes in the positive or negative mental health factors in the control group at T2 and T3.
5. The possible predictors of the training's efficacy were not hypothesized, but examined in exploratory investigations.

Methods:

The final sample was n = 207 with n = 90 in the PoET group and n = 117 in the control. The control group did not receive any intervention in the experimental period, but was offered to participate in a later PoET. The allocation was randomized. Participants in the PoET group completed two online training sessions (3 hours each) via Zoom. Group size was about 25-30 people. The sessions included the following positive psychology constructs: happiness, humour, optimism, loving kindness and gratitude on the first day, and hope, self-efficacy, meaningfulness, forgiveness and resilience on the second day. All participants completed a questionnaire at the beginning of the first training session, at the end of the second one as well as three months after the second session. Participants were given an exercise booklet for all exercises (during the training sessions and at home). The one-week break between the two sessions was advertised as a "7-day-challenge" to improve the motivation in participants to exercise at home.

Data was collected pseudonymised via "qualtrics". Data analyses were conducted with RStudio. For the possible effects of PoET on mental health two-factorial repeated measures ANOVAs were conducted. For the exploration of possible predictors for the efficacy of the training, a hierarchical regression was conducted.

ELIGIBILITY:
Inclusion Criteria:

* legal age (18), ability to use Zoom and all associated technology

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Positive Mental Health Scale (PMH) | before 1st and after 2nd training session, three months after 2nd training session
  9 items, 4-point-scale from 0 ("I do not agree ") to 3 ("I agree"), assessing emotional and psychological aspects of wellbeing, higher scores reflect better positive mental health
Depression Anxiety Stress Scale 21 (DASS-21) | before 1st and after 2nd training session, three months after 2nd training session
  21 items, 4-point-scale from 0 ("did not apply to me at all") to 3 ("applied to me very much or most of the time"), assessing negative emotional states, higher scores reflect more symptoms of depression, anxiety and stress

SECONDARY OUTCOMES:
Life Orientation Test revised (LOT-r) | before 1st and after 2nd training session, three months after 2nd training session
  10 items, 5-point-scale from 0 ("strongly disagree") to 4 ("strongly agree"), assessing dispositional optimism, higher scores reflect higher dispositional optimism
Satisfaction with Life Scale (SWLS) | before 1st and after 2nd training session, three months after 2nd training session
  5 items, 7-point-scale from 1 ("strongly disagree") to 7 ("strongly agree"), assessing global subjective happiness, higher scores indicate a happier person
Brief Resilience Scale (BRS) | before 1st and after 2nd training session, three months after 2nd training session
  6 items, 5-point-scale from 1 ("strongly disagree") to 5 ("strongly agree"), assessing participants' ability to recover from stress despite significant adversity, higher scores reflect higher resilience
Perceived Stress Questionnaire (PSQ) | before 1st and after 2nd training session, three months after 2nd training session
  20 items, 4-point-scale from 1 ("almost never") to 4 ("usually"), assessing the perceived stress in different areas of life, higher scores indicate more stress
Satisfaction in different areas of life | before 1st and after 2nd training session, three months after 2nd training session
  self-generated, five items, 4-point-scale from 1 ("not satisfied") to 4 ("satisfied"), assessing participants satisfaction in five different areas of life, higher scores reflecting higher satisfaction
Implementation of at-home exercices | after 2nd training session and three months after 2nd training session
  self-generated, two questions regarding the frequency and the kind of exercise participants did at home
Socio-demographic data | before 1st training session
  age, gender, marital status, education, employment

CONTACTS AND LOCATIONS:
Overall Officials: Christina Bartnick (born Totzeck), PhD, Study Director — Ruhr-University Bochum
Locations (1):
- Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Niemann L, von Gruner C, Zhang XC, Margraf J, Totzeck C. Positive Emotions Training (PoET) as an online intervention to improve mental health: a feasibility study. BMC Public Health. 2023 Aug 14;23(1):1543. doi: 10.1186/s12889-023-16424-x. PMID 37580658